CLINICAL TRIAL: NCT02034916
Title: A PHASE 2, 2-STAGE, 2-COHORT STUDY OF TALAZOPARIB (BMN 673) ADMINISTERED TO GERMLINE BRCA MUTATION SUBJECTS WITH LOCALLY ADVANCED AND/OR METASTATIC BREAST CANCER
Brief Title: A Phase 2, 2-Stage, 2-Cohort Study of Talazoparib (BMN 673), in Locally Advanced and/or Metastatic Breast Cancer Patients With BRCA Mutation (ABRAZO Study)
Acronym: ABRAZO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary Analysis and study completed. Not stopped due to safety concerns.
Sponsor: Pfizer (Industry)
Collaborators: Myriad Genetic Laboratories, Inc. (Industry); Medivation, Inc. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 673-201; 2013-003076-12 (EudraCT Number); C3441008 (Other: Alias Study Number)
Record Dates: First submitted 2014-01-09; First posted 2014-01-14 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Breast Neoplasms; BRCA 1 Gene Mutation; BRCA 2 Gene Mutation
Keywords: Breast cancer; BRCA mutation; PARP inhibitor; BRCA 1; BRCA 2
MeSH Terms: conditions — Breast Neoplasms | interventions — talazoparib

ARMS (1):
- talazoparib (Experimental): Cohort 1) Subjects with a documented PR or CR to a prior platinum-containing regimen for metastatic disease with disease progression > 8 weeks following the last dose of platinum
  Cohort 2) Subjects who have received > 2 prior chemotherapy regimens for metastatic disease and who have had no prior platinum therapy for metastatic disease
  Interventions: Drug: talazoparib

INTERVENTIONS:
Drug: talazoparib
  Other Names: MDV3800; BMN673

SUMMARY:
The purpose of this 2-stage, 2-cohort Phase 2 trial is to evaluate the safety and efficacy of talazoparib (also known as BMN 673) in subjects with locally advanced or metastatic breast cancer with a deleterious germline BRCA 1 or BRCA 2 mutation. Subjects will be assigned to either Cohort 1 or 2 based on prior chemotherapy for metastatic disease:

* Cohort 1) Subjects with a documented PR or CR to a prior platinum-containing regimen for metastatic disease with disease progression > 8 weeks following the last dose of platinum; or
* Cohort 2) Subjects who have received > 2 prior chemotherapy regimens for metastatic disease and who have had no prior platinum therapy for metastatic disease

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed carcinoma of the breast
* Locally advanced and/or metastatic disease
* Deleterious or pathogenic germline BRCA 1 or BRCA 2 mutation
* Prior chemotherapy: Cohort 1) PR or CR to prior platinum-containing regimen for metastatic disease with disease progression > 8 weeks following the last dose of platinum; or Cohort 2) > 2 prior chemotherapy regimens for metastatic disease and no prior platinum for metastatic disease
* ECOG performance status ≤ 1
* Have adequate organ function

Exclusion Criteria:

* Prior enrollment into a clinical trial of a PARP inhibitor
* CNS metastasis except adequately treated brain metastasis documented by baseline CT or MRI scan that has not progressed since previous scans and that does not require corticosteroids for management of CNS symptoms
* Prior malignancy except for prior BRCA-associated cancer as long as there is no current evidence of the prior cancer, carcinoma in situ of the cervix or non-melanoma skin cancer, and a cancer diagnosed and definitively treated >5 years prior to study enrollment with no subsequent evidence of recurrence
* Known to be HIV positive, active hepatitis C virus, or active hepatitis B virus
* Known hypersensitivity to any of the components of talazoparib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-12-13 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (71):
- United States (37):
  - Marin Cancer Care, Inc., Greenbrae, California
  - UCLA West Medical Pharmacy Attn: Steven L. Wong, PharmD, Los Angeles, California
  - UCLA West Medical Pharmacy, Attn: Steven L. Wong, Pharm.D., Los Angeles, California
  - TRIO-US Central Administration, Los Angeles, California
  - Stanford Women's Cancer Center, Palo Alto, California
  - UCLA Hematology Oncology- Porter Ranch, Porter Ranch, California
  - Torrance Health Association, DBA Torrance Memorial Physician Network/Cancer Care Associates, Redondo Beach, California
  - University of California, San Francisco: Helen Diller Comprehensive Cancer Center, San Francisco, California
  - UCLA Hematology-Oncology, Santa Monica, California
  - Stanford Cancer Institute, Stanford, California
  - Stanford Hospital and Clinics, Stanford, California
  - Sylvester at Deerfield Beach, Deerfield Beach, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - University of Miami Hospital & Clinics, Miami, Florida
  - Memorial Breast Cancer Center at Memorial Hospital West, Pembroke Pines, Florida
  - Memorial Cancer Institute at Memorial Hospital West, Pembroke Pines, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Sylvester at Plantation, Plantation, Florida
  - ICRC, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Investigational Drug Services, Indianapolis, Indiana
  - IU Health University Hospital, Indianapolis, Indiana
  - Sidney & Lois Eskenazi Hospital, Indianapolis, Indiana
  - Springmill Medical Clinic, Indianapolis, Indiana
  - Anne Arundel Medical Center (AAMC), Annapolis Oncology and Hematology, Annapolis, Maryland
  - Anne Arundel Medical Center (AAMC), Research Pharmacy, Annapolis, Maryland
  - Anne Arundel Medical Center (AAMC), Annapolis, Maryland
  - Sidney Kimmel Comprehensive Cancer Center (SKCCC) at Johns Hopkins, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center (SKCCC) at Johns Hopkins, Green Spring Station, Lutherville, Maryland
  - Memorial Sloan Kettering Evelyn H. Lauder Breast Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- France (7):
  - Centre Oscar Lambret, Lille Cédex
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hopital Prive du Confluent, Nantes BP 20215
  - Hopitaux Universitaires de Strasbourg - Hopital Civil, Strasbourg
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse
  - CHU Bretonneau Centre Henry Kaplan, Tours
- Germany (12):
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - IOZ Muenchen - lnerdisziplinaeres Onkologisches Zentrum, Munich, Bavaria
  - University of Munich (LMU) Grosshadern Hospital, Munich, Bavaria
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Klinikum Mutterhaus Der Borromaeerinnen Ggmbh, Trier, Rhineland-Palatinate
  - University Hospital Carl Gustav Carus, Dresden, Saxony
  - Helios Klinikum Berlin-Buch, Berlin
  - University Hospital Duesseldorf, Düsseldorf
  - Kliniken Essen Mitte Klinik fuer Gynaekologie und Gynaekologische Onkologie, Essen
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - g.SUND Gynaekologie Kompetenzzentrum Stralsund, Stralsund
  - Universitaets-Frauenklinik, Tübingen
- Spain (9):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital General Universitario Gregorio Maranon, Madrid
  - MD Anderson Cancer Center International Espana, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario San Juan de Alicante, Sant Joan d'Alacant
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (6):
  - Cambridge University Hospital NHS Foundation Trust, Cambridge, England
  - Sarah Cannon Research Institute UK, London, England
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston, Lancashire
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Turner NC, Laird AD, Telli ML, Rugo HS, Mailliez A, Ettl J, Grischke EM, Mina LA, Balmana J, Fasching PA, Hurvitz SA, Hopkins JF, Albacker LA, Chelliserry J, Chen Y, Conte U, Wardley AM, Robson ME. Genomic analysis of advanced breast cancer tumors from talazoparib-treated gBRCA1/2mut carriers in the ABRAZO study. NPJ Breast Cancer. 2023 Oct 6;9(1):81. doi: 10.1038/s41523-023-00561-y. PMID 37803017
- [Derived] Turner NC, Telli ML, Rugo HS, Mailliez A, Ettl J, Grischke EM, Mina LA, Balmana J, Fasching PA, Hurvitz SA, Wardley AM, Chappey C, Hannah AL, Robson ME; ABRAZO Study Group. A Phase II Study of Talazoparib after Platinum or Cytotoxic Nonplatinum Regimens in Patients with Advanced Breast Cancer and Germline BRCA1/2 Mutations (ABRAZO). Clin Cancer Res. 2019 May 1;25(9):2717-2724. doi: 10.1158/1078-0432.CCR-18-1891. Epub 2018 Dec 18. PMID 30563931

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, enrollment of participants was to be done in 2 stages for each of the 2 cohorts. Sufficient responses in each cohort were observed such that enrollment could proceed to Stage 2 for both cohorts. However, due to Sponsor decision, enrollment in the overall trial was terminated early.
Groups:
- Cohort 1: Talazoparib 1 mg: Participants who responded to a prior platinum-containing treatment for metastatic breast cancer, with disease progression of at least 8 weeks following the last dose of platinum, received talazoparib 1.0 milligram (mg) orally, once daily for 21 days in repeated 21-day cycles until disease progression, occurrence of unacceptable toxicity or permanent treatment discontinuation. Participants were followed-up for survival and new anticancer treatment at every 60 days after the last dose of study drug for the first year, every 90 days thereafter.
- Cohort 2: Talazoparib 1 mg: Participants with more than 2 prior non-platinum chemotherapy treatment for metastatic breast cancer, received talazoparib 1.0 mg orally, once daily for 21 days in repeated 21-day cycles until disease progression, occurrence of unacceptable toxicity or permanent treatment discontinuation. Prior adjuvant or neo-adjuvant therapy with a platinum was allowed if first disease recurrence was for more than 6 months since last dose of adjuvant/neo-adjuvant platinum treatment. Participants were followed-up for survival and new anticancer treatment at every 60 days after the last dose of study drug for the first year, every 90 days thereafter.
Period: Overall Study
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Started | 49 | 35
Treated | 48 | 35
Completed | 0 | 0
Not Completed | 49 | 35
Not completed — Death | 39 | 28
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 4 | 1
Not completed — Study terminated by sponsor | 4 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population involved all enrolled participants including participants who were not treated.
Groups:
- Cohort 1: Talazoparib 1 mg: Participants who responded to a prior platinum-containing treatment for metastatic breast cancer, with disease progression of at least 8 weeks following the last dose of platinum, received talazoparib 1.0 mg orally, once daily for 21 days in repeated 21-day cycles until disease progression, occurrence of unacceptable toxicity or permanent treatment discontinuation. Participants were followed-up for survival and new anticancer treatment at every 60 days after the last dose of study drug for the first year, every 90 days thereafter.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg | Total
Number analyzed (Participants) | 49 | 35 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (11.48) | 53.4 (11.05) | 51.5 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 34 | 82
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR: Percentage of participants with a confirmed best overall complete response (CR) or partial response (PR) according to response evaluation criteria in solid tumors version 1.1 (RECIST 1.1). CR: Disappearance of all non-nodal target and non-target lesions, including target and non-target lymph nodes reduction to less than (<) 10 millimeter (mm) in short axis. PR: Greater than or equal to (>=) 30 percent (%) decrease in sum of diameters of target lesions, compared to the sum at baseline. Response evaluation was done by an independent radiology facility (IRF).
Time Frame: From randomization until data cutoff date (01 Sep 2016)
Population: Tumor-evaluable population (TEP) included all treated participants who had a baseline and at least 1 post-baseline tumor assessment or who discontinued the study before first scheduled post-baseline tumor scan plus (+) 1 week window.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 48 | 35
percentage of participants | 20.8 [10.47 to 34.99] | 37.1 [21.47 to 55.08]

2. Secondary Outcome: Clinical Benefit Rate-24 (CBR-24)
Description: CBR24: Percentage of participants with a best response of CR, PR or stable disease (SD) sustained for at least 24 weeks, as assessed by IRF using RECIST 1.1. CR: Disappearance of all non-nodal target and non-target lesions, including target and non-target lymph nodes reduction to <10 mm in short axis. PR: >=30% decrease in sum of diameters of target lesions, compared to the sum at baseline. SD: Neither PR nor progression of disease (PD) criteria met. SD follow PR only when sum increases by less than 20% from the nadir, but previously seen 30% decrease from baseline no longer hold. PD: >=20% increase (>=5 mm absolute increase) in the sum of target lesion measurements, compared to the smallest sum on study (including baseline), or unequivocal progression of non-target lesions, evaluated as a whole, such that it is clear that treatment has failed and disease is progressing, regardless of the status of the target lesions.
Time Frame: From randomization until data cutoff date (01 Sep 2016)
Population: TEP included all treated participants who had a baseline and at least 1 post-baseline tumor assessment or who discontinued the study before first scheduled post-baseline tumor scan + 1 week window.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 48 | 35
percentage of participants | 27.1 [15.28 to 41.85] | 45.7 [28.83 to 63.35]

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR: Time from first documentation of CR or PR, to PD by IRF assessment using RECIST 1.1, or to death due to any cause, whichever occurred first. CR: Disappearance of all non-nodal target and non-target lesions, with target and non-target lymph nodes reduction to <10 mm in short axis. PR: >=30% decrease in sum of diameters of target lesions, compared to the sum at baseline. PD: >=20% increase (>=5 mm absolute increase) in the sum of target lesion measurements, compared to the smallest sum on study (including baseline), or unequivocal progression of non-target lesions, evaluated as a whole, such that it is clear that treatment has failed and disease is progressing, regardless of the status of the target lesions. Participants with no PD or death at the analysis date were censored at last tumor assessment date prior to on or before initiation of a new anticancer therapy or before the data cutoff date.
Time Frame: From first documentation of CR or PR until PD, last tumor assessment without PD before new anticancer treatment initiation or death due to any cause, whichever occurred first (up to the data cutoff date [01 Sep 2016])
Population: TEP included all treated participants who had a baseline and at least 1 post-baseline tumor assessment or who discontinued the study before first scheduled post-baseline tumor scan + 1 week window. Here 'Number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 10 | 13
months | 5.8 [2.8 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient number of events at the time of data cutoff (01 Sep 2016). | 3.8 [2.8 to 10.1]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time in months from the first dose of study drug to the first documentation of PD by investigator assessment using RECIST 1.1 or death on study due to any cause on or before the data cutoff date, whichever occurred first. PD: >=20% increase (>=5 mm absolute increase) in the sum of target lesion measurements, compared to the smallest sum on study (including baseline), or unequivocal progression of non-target lesions, evaluated as a whole, such that it is clear that treatment has failed and disease is progressing, regardless of the status of the target lesions. Participants with no PFS event at the analysis were censored at last tumor assessment date prior to data cutoff or date of new anticancer treatment initiation, whichever occurred first.
Time Frame: From first dose of study drug until PD, last tumor assessment without PD before new anticancer treatment initiation or death due to any cause, whichever occurred first (up to the data cutoff date [01 Sep 2016])
Population: ITT population involved all enrolled participants including participants who were not treated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 49 | 35
months | 4.0 [2.8 to 5.4] | 5.6 [5.5 to 7.8]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of study drug to death due to any cause. For participants without a death date at the time of data cutoff or permanently lost to follow-up, OS was right-censored at the date the participant was last known to be alive on or before the data cutoff date.
Time Frame: From first dose of study drug until death due to any cause (up to the data cutoff date [01 Sep 2016])
Population: ITT population involved all enrolled participants including participants who were not treated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 49 | 35
months | 11.8 [8.8 to 15.0] | 16.5 [10.1 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient number of events at the time of data cutoff (01 Sep 2016).

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; an important medical event or reaction, including events requiring medical intervention to prevent worsening to any of the previously noted seriousness criteria. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious AEs.
Time Frame: Baseline up to end of study (up to a maximum duration of 42.8 months): based on data cutoff date (31 Oct 2018)
Population: Safety population included all participants who received at least 1 dose of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 48 | 35
Participants
  AEs | 47 [8.8 to 15.0] | 34 [10.1 to NA]
  SAEs | 16 | 7

7. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: A treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. A treatment-related SAE was a treatment-related AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; an important medical event or reaction, including events requiring medical intervention to prevent worsening to any of the previously noted seriousness criteria. Related TEAEs are TEAEs that were judged by the investigators as possibly, probably, or definitely related to study drug. AEs included both SAES and non SAES.
Time Frame: Baseline up to end of study (up to a maximum duration of 42.8 months): based on data cutoff date (31 Oct 2018)
Population: Safety population included all participants who received at least 1 dose of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 48 | 35
Participants
  AEs | 46 | 33
  SAEs | 7 | 4

8. Secondary Outcome: Number of Participants With Outcome in Response to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Outcome of an AE was response to a question answered by the investigator: 'Is the AE leading to study discontinuation or death?' as 'yes'.
Time Frame: Baseline up to end of study (up to a maximum duration of 42.8 months): based on data cutoff date (31 Oct 2018)
Population: Safety population included all participants who received at least 1 dose of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 48 | 35
Participants
  AEs leading to study drug discontinuation | 4 | 1
  AEs leading to death | 5 | 1

9. Secondary Outcome: Number of Participants With Toxicity Grades Increase of 2 or More in Laboratory Parameter (Hematology Parameter)
Description: Laboratory tests included hematology (hemoglobin [low], leucocytes [low], lymphocytes [low], neutrophils [low], platelets [low]). Toxicity grades were evaluated based on national cancer institute- common terminology criteria for adverse events (NCI-CTCAE) version 4.03. Number of participants with increase of 2 or more CTCAE toxicity grades above baseline, for hematology laboratory parameter is reported in this outcome measure.
Time Frame: Baseline up to end of study (up to a maximum duration of 42.8 months): based on data cutoff date (31 Oct 2018)
Population: Safety population included all participants who received at least 1 dose of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 48 | 35
Participants
  Hemoglobin (low) | 19 | 16
  Leukocytes (low) | 16 | 15
  Lymphocytes (low) | 15 | 4
  Neutrophils (low) | 20 | 17
  Platelets (low) | 21 | 10

10. Secondary Outcome: Number of Participants With Toxicity Grades Increase of 2 or More in Laboratory Parameter (Chemistry Parameter)
Description: Laboratory tests included serum chemistry (alanine aminotransferase [high], albumin [low], alkaline phosphatase [high], aspartate aminotransferase [high], bilirubin [high], calcium [low], glucose [high], magnesium [low], phosphate [low], potassium [high], potassium [low], sodium [high], sodium [low]). Toxicity grades were evaluated based on national cancer institute- common terminology criteria for adverse events (NCI-CTCAE) version 4.03. Number of participants with increase of 2 or more CTCAE toxicity grades above baseline, for chemistry laboratory parameter is reported in this outcome measure.
Time Frame: Baseline up to 30 days after the last dose of study drug or before initiation of a new anticancer treatment, whichever occurred first (up to data cutoff date [01 Sep 2016])
Population: Safety population included all participants who received at least 1 dose of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 48 | 35
Participants
  Alanine aminotransferase (high) | 3 | 2
  Albumin (low) | 3 | 0
  Alkaline phosphatase (high) | 1 | 1
  Aspartate aminotransferase (high) | 2 | 1
  Bilirubin (high) | 2 | 0
  Calcium (low) | 4 | 1
  Glucose (high) | 1 | 1
  Magnesium (low) | 1 | 0
  Phosphate (low) | 6 | 2
  Potassium (high) | 1 | 0
  Potassium (low) | 2 | 0
  Sodium (high) | 1 | 0
  Sodium (low) | 0 | 1

11. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Criteria for clinically significant vital signs changes: 1) Blood pressure: systolic blood pressure (SBP): greater than or equal to (>=30) millimeters of mercury (mmHg) increase from baseline, diastolic blood pressure (DBP): >=20 mmHg decrease from baseline; 2) Heart rate (HR): absolute HR greater than (>) 120 beats per minute (bpm) and >30 bpm increase from baseline, absolute HR less than (<) 50 bpm and >20 bpm decrease from baseline; 3) Weight: >10% decrease from baseline. Number of participants with any clinically significant change from baseline for blood pressure, heart rate and weight are reported in this outcome measure.
Time Frame: Baseline up to end of study (up to a maximum duration of 42.8 months): based on data cutoff date (31 Oct 2018)
Population: Safety population included all participants who received at least 1 dose of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 48 | 35
Participants
  Blood pressure (SBP or DBP) | 20 | 18
  HR | 2 | 0
  Weight | 4 | 1

12. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Findings
Description: Physical examination included examination of the head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The examination assessed the participants for any potential changes in general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms. Findings were considered to be clinically significant based on investigator's decision.
Time Frame: Baseline up to end of study (up to a maximum duration of 42.8 months): based on data cutoff date (31 Oct 2018)
Population: Safety population included all participants who received at least 1 dose of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 48 | 35
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With At Least 1 Concomitant Medication
Description: Number of participants taking any non-study medications, therapies, including herbal supplements during the treatment-emergent period for the management of an adverse event or for the treatment of any other disease.
Time Frame: Baseline up to end of study (up to a maximum duration of 42.8 months): based on data cutoff date (31 Oct 2018)
Population: Safety population included all participants who received at least 1 dose of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 48 | 35
Participants | 48 | 34

14. Secondary Outcome: Trough Concentration Versus Time Summary of Talazoparib
Description: Concentrations below the limit of quantitation values less than or equal to (<=) 25 picogram per milliliter (pg/mL) were set as zero. Pharmacokinetic (PK) analysis was not done separately for each reporting arm and cohorts were combined for PK analysis.
Time Frame: Predose on Day 1 of Cycle 1, 2, 3, and 4 (data cutoff date: 01 Sep 2016)
Population: PK population included all participants who received at least 1 dose of talazoparib and had evaluable PK assessments. Here 'n' signifies participants evaluable for each specified categories.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Cohort 1 + Cohort 2: Talazoparib 1 mg: Participants, who either responded to a prior platinum-containing treatment for metastatic breast cancer or had more than 2 prior non-platinum chemotherapy treatment for metastatic breast cancer, received talazoparib 1.0 mg orally, once daily for 21 days in repeated 21-day cycles until disease progression, occurrence of unacceptable toxicity or permanent treatment discontinuation. For the participants with non-platinum chemotherapy, prior adjuvant or neo-adjuvant therapy with a platinum was allowed if first disease recurrence was for more than 6 months since last dose of adjuvant/neo-adjuvant platinum treatment. Participants were followed-up for survival and new anticancer treatment at every 60 days after the last dose of study drug for the first year, every 90 days thereafter.
Arm/Group | Cohort 1 + Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 83
pg/mL
  Day 1 of Cycle 1: number analyzed (Participants) | 82
  Day 1 of Cycle 1 | 10.3 (93.3)
  Day 1 of Cycle 2: number analyzed (Participants) | 63
  Day 1 of Cycle 2 | 4340 (2360)
  Day 1 of Cycle 3: number analyzed (Participants) | 44
  Day 1 of Cycle 3 | 4510 (2720)
  Day 1 of Cycle 4: number analyzed (Participants) | 33
  Day 1 of Cycle 4 | 3660 (1690)

15. Other Pre Specified Outcome: Time to Deterioration in Global Health Status/Quality of Life (QOL) and Functional Status as Assessed by European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30)
Description: Time to deterioration was defined as the time from baseline to day to death, first occurrence of progression, or a >=10 point change from baseline in any of the functional status score and global health status/QOL score based on the EORTC-QLQ-C30, whichever occurred first. EORTC-QLQ-C30 questionnaire is a standardized instrument developed to assess the quality of life of people with cancer. EORTC-QLQ-C30 functional subscale includes 5 items: physical, role, emotional, cognitive, and social functioning. All of the single items of functional status subscale measures and global health status/QOL subscale range from 0 to 100, where higher scores represent a better level of functioning/quality of life.
Time Frame: Baseline up to death, disease progression or end of treatment (30 days after last dose of study drug or before initiation of a new anticancer therapy, whichever occurred first [up to data cutoff date: 01 Sep 2016])
Population: ITT population involved all enrolled participants including participants who were not treated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 49 | 35
months
  Global Health Status/QOL | 2.8 (18.33) [2.1 to 3.0] | 5.5 (32.81) [4.2 to 5.7]
  Physical Functioning | 3.1 (15.84) [2.1 to 4.6] | 5.6 (21.60) [5.3 to 7.7]
  Role Functioning | 2.1 (15.43) [1.4 to 2.8] | 4.2 (31.67) [2.1 to 5.5]
  Emotional Functioning | 2.7 (19.29) [2.0 to 2.8] | 5.5 (24.45) [4.3 to 5.6]
  Cognitive Functioning | 2.7 (21.36) [1.6 to 3.2] | 4.2 (15.47) [2.8 to 5.5]
  Social Functioning | 2.2 (19.42) [1.4 to 2.9] | 5.3 (23.57) [4.1 to 5.6]

16. Other Pre Specified Outcome: Time to Deterioration in Disease Specific Symptoms as Assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Breast Cancer Module (EORTC-QLQ-BR23)
Description: Time to deterioration was defined as the time from baseline to day to death, first occurrence of progression, or a >=10 point change from baseline in any of the symptom score based on the EORTC-QLQ-BR23, whichever occurred first. EORTC-QLQ-BR23 is a disease-specific module for breast cancer developed as a supplement for the EORTC-QLQ-C30 to assess the quality of life of participants with breast cancer. EORTC-QLQ-BR23 symptoms subscale includes 4 items: systemic therapy side effects, breast symptoms, arm symptoms, upset by hair loss. Each item is rated by choosing 1 of 4 possible responses that record the level of intensity (1= not at all, 2= a little, 3= quite a bit, and 4= very much) within each scale.
Time Frame: as for outcome 15
Population: ITT population involved all enrolled participants including participants who were not treated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Number analyzed (Participants) | 49 | 35
months
  Systemic Therapy Side Effects | 2.8 (5.69) [2.3 to 4.0] | 5.5 (11.93) [4.1 to 5.6]
  Breast Symptoms | 3.1 (9.71) [2.5 to 4.6] | 5.6 (28.50) [5.3 to 7.7]
  Arm Symptoms | 2.6 (8.27) [2.0 to 3.7] | 4.2 (8.07) [2.8 to 5.5]
  Upset by Hair Loss | 4.0 [2.7 to 5.4] | 5.6 [5.3 to 7.7]

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (up to maximum duration of 42.8 months)
Description: Same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. AEs and SAEs were collected for safety population.
Arm/Group | Cohort 1: Talazoparib 1 mg | Cohort 2: Talazoparib 1 mg
Serious Adverse Events (participants affected / at risk) | 16/48 | 7/35
Other Adverse Events (participants affected / at risk) | 47/48 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cohort 1: Talazoparib 1 mg (N=48) | Cohort 2: Talazoparib 1 mg (N=35)
Anaemia (Blood and lymphatic system disorders) | 5 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Silicon granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lipoinjection (Surgical and medical procedures) | 1 | 0
Salpingo-oophorectomy (Surgical and medical procedures) | 1/47 | 0/34 — Gender specific event.
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Talazoparib 1 mg (N=48) | Cohort 2: Talazoparib 1 mg (N=35)
Anaemia (Blood and lymphatic system disorders) | 23 | 19
Leukopenia (Blood and lymphatic system disorders) | 7 | 6
Lymphopenia (Blood and lymphatic system disorders) | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 10 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 9
Tachycardia (Cardiac disorders) | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 7 | 7
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6
Constipation (Gastrointestinal disorders) | 9 | 6
Diarrhoea (Gastrointestinal disorders) | 18 | 10
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 20 | 15
Stomatitis (Gastrointestinal disorders) | 3 | 1
Toothache (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 10 | 8
Asthenia (General disorders) | 3 | 10
Axillary pain (General disorders) | 1 | 2
Fatigue (General disorders) | 29 | 8
Mucosal inflammation (General disorders) | 4 | 2
Non-cardiac chest pain (General disorders) | 3 | 0
Oedema peripheral (General disorders) | 1 | 6
Pyrexia (General disorders) | 1 | 5
Gingivitis (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 3 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 3
Rhinitis (Infections and infestations) | 4 | 2
Sinusitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 5
Alanine aminotransferase increased (Investigations) | 1 | 3
Aspartate aminotransferase increased (Investigations) | 4 | 2
Neutrophil count decreased (Investigations) | 5 | 5
Platelet count decreased (Investigations) | 7 | 5
Weight decreased (Investigations) | 3 | 0
White blood cell count decreased (Investigations) | 3 | 5
Decreased appetite (Metabolism and nutrition disorders) | 12 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Dizziness (Nervous system disorders) | 6 | 2
Dysgeusia (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 9 | 11
Neuralgia (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 4
Depression (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Hot flush (Vascular disorders) | 3 | 3
Lymphoedema (Vascular disorders) | 3 | 2
Chills (General disorders) | 1 | 2
Oral herpes (Infections and infestations) | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 11 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Presyncope (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.